CLINICAL TRIAL: NCT02634268
Title: INtervention Study In overweiGHT Patients With COPD
Acronym: INSIGHT COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1U01HL128868 (NIH)
Record Dates: First submitted 2015-12-10; First posted 2015-12-18 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Obesity; Weight Loss; Life Style; Overweight
Keywords: randomized controlled trial; diet; exercise; obesity; overweight; chronic obstructive pulmonary disease; lifestyle
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity; Weight Loss; Overweight; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle intervention (Active Comparator): Behavioral lifestyle intervention focused on healthy eating and physical activity
  Interventions: Behavioral: Lifestyle Intervention
- Usual Care (No Intervention): Participants continue with usual diet and exercise activities as they desire

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Behavioral lifestyle intervention focused on healthy eating and physical activity
  Arms: Lifestyle intervention

SUMMARY:
Symptoms of chronic obstructive pulmonary disease (COPD) and high body mass index (BMI) overlap. The investigators are trying to find out if a program proven to help people lose a modest amount of weight and increase their physical activity will improve COPD symptoms for those with a high BMI. The program uses a series of video sessions and self-study handouts focused on healthy eating and increasing physical activity, and encourages participants to monitor their weight, diet, and physical activity for one year. For those who want to, they will be able to work with a health coach to help meet weight and activity goals. We hope that the program will lead to improved exercise tolerance, body weight, dyspnea, generic health-related quality of life, and major cardiovascular risk factors (central obesity by waist circumference, Framingham Risk Score, and blood pressure) through 12 months of follow-up. To be in the study, participants will need to have COPD, high BMI, history of smoking, shortness of breath, and be at least 40 years old.

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older at time of eligibility screening;
* Body mass index 25.0-44.9 kg/m2 (also see Figure 2);
* Smoked more than 10 pack-years of cigarettes;
* Shortness of breath;
* COPD;
* Able to participate fully in all study protocol/procedures including written informed consent process.

Exclusion Criteria:

* Inability to speak, read, or understand English;
* Active weight loss interventions;
* Expected weight loss because of alternate explanations, such as from illness;
* Unable to ambulate to weight scale for weight measurement;
* Safety and/or adherence concerns due to severe physical or mental health issues or life expectancy <18 months;
* Pregnant, lactating, or planning to become pregnant during the study period;
* Participation in other intervention studies.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Au, MD, MS, Principal Investigator — VA Puget Sound Health Care System; Jun Ma, MD, PhD, Principal Investigator — University of Illinois at Chicago - Institute for Health Research and Policy
Locations (39):
- United States (39):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - University of Alabama at Birmingham - UAB Lung Health Center, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - Universtiy of California, San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Waterbury Pulmonary Associates, Waterbury, Connecticut
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Northwestern University - Northwestern Medical Group - Pulmonology, Chicago, Illinois
  - University of Illinois, Chicago - Division of Pulmonay, Critical Care, Sleep & Allergy, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Chest Medicine, South Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University - Pulmonary & Critical Care Medicine, Baltimore, Maryland
  - Boston VA Medical Center, Boston, Massachusetts
  - Baystate Health, Springfield, Massachusetts
  - University of Michigan - Division of Pulmonary & Critical Care Medicine, Ann Arbor, Michigan
  - Minneapolis VA Health Care System - Pulmonology, Minneapolis, Minnesota
  - Minnesota Health Partners, Saint Paul, Minnesota
  - St. Louis VA, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - University of Buffalo, Buffalo, New York
  - Buffalo VA Medical Center, Buffalo, New York
  - NYU Winthrop, Mineola, New York
  - Duke University, Durham, North Carolina
  - East Carolina University - Pulmonary, Critical Care & Sleep Medicine, Greenville, North Carolina
  - Case Western, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S. Hershey Medical Center - Pulmonary, Allergy & Critical Care Medicine, Hershey, Pennsylvania
  - Temple University Hospital - Temple Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Kaufmann Building, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - BSW Research, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Grand Medical Clinic, Katy, Texas
  - University of Utah, Salt Lake City, Utah
  - White River Junction VA, White River Junction, Vermont
  - VA Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be shared with NHLBI's data repository, Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Summer 2022 and onward according to BioLINCC policy.
Access Criteria: Researchers may submit a data request vis BioLINCC, including description of the research plan/protocol, and documentation of review from an Institutional Review Board (IRB) or Ethics Committee (EC). Once those requirements are met and the request is approved by the NHLBI, BioLINCC staff will provide a Research Materials Distribution Agreement (RMDA) to be signed by a designated Principal Investigator and an authorized business official from the receiving institution, prior to data release.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Derived] Au DH, Gleason E, Hunter-Merrill R, Baron AE, Collins M, Ronneberg C, Lv N, Rise P, Wai TH, Plumley R, Wisniewski SR, Sciurba FC, Kim DY, Simonelli P, Krishnan JA, Wendt CH, Feemster LC, Criner GJ, Maddipati V, Mohan A, Ma J. Lifestyle Intervention and Excess Weight in Chronic Obstructive Pulmonary Disease (COPD): INSIGHT COPD Randomized Clinical Trial. Ann Am Thorac Soc. 2023 Dec;20(12):1743-1751. doi: 10.1513/AnnalsATS.202305-458OC. PMID 37769182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 4/28/2017-8/16/2019 from 38 diverse settings across the United States, including rural, urban, and academic medical centers, and Department of Veteran Affairs Health Systems.
Period: Overall Study
Arm/Group | Lifestyle Intervention | Usual Care
Started | 346 | 338
Completed | 287 (In-person visit completion = 267 for both groups. Some participants completed only surveys because of Covid-19 restrictions.) | 291 (In-person visit completion = 267 for both groups. Some participants completed only surveys because of Covid-19 restrictions.)
Not Completed | 59 | 47

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Intervention | Usual Care | Total
Number analyzed (Participants) | 346 | 338 | 684
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (8.2) | 66.9 (7.7) | 67.0 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 140 | 282
  Male | 204 | 198 | 402
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 337 | 333 | 670
  Unknown or Not Reported | 5 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 67 | 69 | 136
  White | 267 | 260 | 527
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Six Minute Walk Test
Description: distance walked in six minutes
Time Frame: 12 months
Population: We report here the unadjusted means at 12 months. The analysis population for adjusted between-group difference includes study participants with a measurement at baseline and/or 12 months; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
feet | 1071.0 (354.1) | 1005.9 (339.0)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12-month six minute walk test distance between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = .02, Mixed Models Analysis; Difference in average six minute walk test distance at 12 months between control and intervention groups; Mean Difference (Final Values) = 42.3, 95% CI 2-sided [7.93 to 76.6] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

2. Secondary Outcome: Modified Borg Scale
Description: Shortness of breath: scores range from 0 (nothing at all) to 10 (very, very severe).
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
units on a scale | 2.7 (1.9) | 3.2 (1.9)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12-month Modified Borg Scale score between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = .0008, Mixed Models Analysis; Difference in average Modified Borg Scale score at 12 months between control and intervention groups; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.63 to -0.09] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

3. Secondary Outcome: Weight
Description: body weight
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
kilograms | 91.0 (17.7) | 93.7 (17.0)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12-month body weight between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Difference in average body weight at 12 months between control and intervention groups; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-2.33 to -0.34] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

4. Secondary Outcome: Short Form 12 Health Survey (SF-12) Physical Component Score (PCS)
Description: scores range from 0-100 with higher scores reflecting better health
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
score on a scale | 39.7 (8.5) | 37.5 (8.8)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12-month SF-12 PCS between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = 0.01, Mixed Models Analysis; Difference in average SF-12 PCS at 12 months between control and intervention groups; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [0.35 to 2.60] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

5. Secondary Outcome: Short Form 12 Health Survey (SF-12) Mental Component Score (MCS)
Description: scores range from 0-100 with higher scores reflecting better health
Time Frame: 12-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
score on a scale | 51.7 (9.7) | 51.4 (9.8)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12-month SF-12 MCS between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = 0.45, Mixed Models Analysis; Difference in average SF-12 MCS at 12 months between control and intervention groups; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-0.84 to 1.89] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

6. Secondary Outcome: Non-laboratory Framingham Risk Score
Description: This measure uses non-laboratory-based measures (sex, age, body mass index, systolic blood pressure, use of antihypertensive treatment, smoking status, and diabetes status) to yield a score (cardiovascular disease points) representing 10-year risk of having a cardiovascular problem. Low scores (minimum of -2 for women, -3 for men) indicate low risk. Scores of 21 or higher indicate high risk (30% risk or higher).
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 345 | 338
score on a scale | 15.0 (3.0) | 15.4 (3.0)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12-month Framingham Risk Score between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = 0.009, Mixed Models Analysis; Difference in average Framingham Risk Score at 12 months between control and intervention groups; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.71 to -0.10]

7. Secondary Outcome: Waist Circumference
Description: cardiovascular disease risk
Time Frame: 12 months
Population: We report here the unadjusted means at 12 months. The analysis population for adjusted between-group difference includes study participants with a measurement at baseline and/or 12-months; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
centimeters | 111.3 (12.9) | 113.1 (13.5)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12 month waist circumference between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = 0.13, Mixed Models Analysis; Difference in average waist circumference at 12 months between control and intervention groups; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-2.12 to 0.26] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

8. Secondary Outcome: Systolic Blood Pressure
Description: indicator of cardiovascular disease risk; higher values indicate higher risk
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
mmHg | 129.5 (17.2) | 128.8 (16.2)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12-month systolic blood pressure between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = 0.64, Mixed Models Analysis; Difference in average 12 month systolic blood at 12 months between control and intervention groups; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-3.02 to 1.84] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

9. Secondary Outcome: Body Mass Index (BMI)
Description: cardiovascular disease risk
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
kg/m^2 | 31.9 (5.0) | 32.7 (4.8)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12-month BMI between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = 0.004, Mixed Models Analysis; Difference in average BMI at 12 months between control and intervention groups; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.85 to -0.17] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

10. Secondary Outcome: St George's Respiratory Questionnaire For COPD Patients (SGRQ-C) Symptom Component Score
Description: Designed to measure respiratory health quality of life in patients with COPD, providing a total score and three subscale scores assessing: (1) symptoms (frequency and severity), (2) activities that cause or are limited by breathlessness and (3) Impact (social functioning and psychological disturbances resulting from COPD). Each score ranges from 0-100, with higher scores indicating more limitations.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
score on a scale | 52.6 (21.9) | 54.9 (20.8)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12 month SGRQ-C Symptom score between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = 0.09, Mixed Models Analysis; Difference in average SGRQ-C Symptom score at 12 months between control and intervention groups; Mean Difference (Final Values) = -2.25, 95% CI 2-sided [-4.87 to 0.36]; Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

11. Secondary Outcome: St George's Respiratory Questionnaire For COPD Patients (SGRQ-C) Activity Component Score
Description: as for outcome 10
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
score on a scale | 58.9 (25.8) | 63.3 (25.3)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12 month SGRQ-C Activity score between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = 0.12, Mixed Models Analysis; Difference in average SGRQ-C Activity score at 12 months between control and intervention groups; Mean Difference (Final Values) = -2.31, 95% CI 2-sided [-5.19 to 0.56] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

12. Secondary Outcome: St George's Respiratory Questionnaire For COPD Patients (SGRQ-C) Impact Component Score
Description: as for outcome 10
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
score on a scale | 29.2 (20.1) | 32.8 (21.5)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12 month SGRQ-C Impact score between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = 0.03, Mixed Models Analysis; Difference in average SGRQ-C Impact score at 12 months between control and intervention groups; Mean Difference (Final Values) = -2.72, 95% CI 2-sided [-5.19 to -0.25] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

13. Secondary Outcome: St George's Respiratory Questionnaire For COPD Patients (SGRQ-C) Total Score
Description: as for outcome 10
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 346 | 338
score on a scale | 42.4 (19.5) | 46.1 (19.8)
Statistical Analysis 1: Comparison: Lifestyle Intervention vs Usual Care; Linear mixed model analysis, including participants with a measurement at baseline and/or 12 months, comparing the average 12-month SGRQ-C Total score between control and intervention groups. Our analysis controlled for smoking and before/during the COVID-19 pandemic with fixed effects, while random effects were used for multiple measurement on individuals and study sites; Test type: Superiority; p = 0.03, Mixed Models Analysis; Difference in average SGRQ-C Total score at 12 months between control and intervention groups; Mean Difference (Final Values) = -2.42, 95% CI 2-sided [-4.55 to -0.28] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

ADVERSE EVENTS:
Time Frame: We systematically collected adverse events (AE) by body system at the 12-month visit. Lifestyle coaches also learned about AEs through their interaction with participants.
Description: Adverse events were monitored without regard to the specific Adverse Event Term.
Arm/Group | Lifestyle Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 4/346 | 9/338
Serious Adverse Events (participants affected / at risk) | 78/346 | 75/338
Other Adverse Events (participants affected / at risk) | 95/346 | 90/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Intervention (N=346) | Usual Care (N=338)
Cardiovascular (General disorders) | 22 (27) | 20 (27)
Dermatological (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5)
Gastrointestinal (Gastrointestinal disorders) | 14 (16) | 7 (9)
Hematological (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Metabolic (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (7)
Neurological (Nervous system disorders) | 7 (7) | 7 (8)
Psychological (Psychiatric disorders) | 2 (4) | 2 (2)
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 35 (42) | 35 (50)
Renal/Urologic (Renal and urinary disorders) | 7 (9) | 11 (11)
Hepatobiliary (Hepatobiliary disorders) | 4 (4) | 3 (3)
Other (General disorders) | 13 (14) | 14 (14)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Intervention (N=346) | Usual Care (N=338)
Cardiovascular (General disorders) | 20 (21) | 14 (16)
Dermatological (Skin and subcutaneous tissue disorders) | 12 (15) | 11 (12)
Gastrointestinal (Gastrointestinal disorders) | 6 (6) | 10 (13)
Hematological (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Metabolic (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 30 (35) | 24 (29)
Neurological (Nervous system disorders) | 7 (8) | 6 (7)
Psychological (Psychiatric disorders) | 4 (5) | 3 (4)
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 38 (47) | 52 (67)
Renal/Urologic (Renal and urinary disorders) | 3 (4) | 5 (5)
Hepatobiliary (Hepatobiliary disorders) | 0 (0) | 2 (2)
Other (General disorders) | 16 (19) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT02634268/Prot_SAP_000.pdf